CLINICAL TRIAL: NCT01949259
Title: Rapid Learning in Practice: A Lung Cancer Survival Decision Support System in Routine Patient Care Data
Brief Title: Rapid Learning for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Liverpool Cancer Therapy Centre (Other Government); Macarthur Cancer Therapy Centre, Liverpool (Other); Ingham Institute Hospital, Liverpool (Unknown); NSW, Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: Rapid learning lung cancer
Record Dates: First submitted 2013-09-10; First posted 2013-09-24 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: Retrospective; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective collection: Retrospective collection of data from included lung cancer patients.

SUMMARY:
A retrospective, data mining project that re-uses routine patient care data for decision support systems.

DETAILED DESCRIPTION:
By installing tools that extract clinical data from electronic health records and image data from the Picture Archiving and Communication System, decision support systems are built and validated that can predict survival and treatment toxicities of lung cancer patients treated with radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Patients notes as suffering from lung cancer in at least one clinical data source.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Survival | From radiotherapy until death
  Retrospective data will be collected from each included patient from start of radiotherapy until end of study or death (an expected average of 10 years).

SECONDARY OUTCOMES:
Local control | From start of treatment until death,
  Data will be collected from inclusion in the study until end of study of death (an expected average time frame of 10 years) concerning the local control of this tumour.
Distant metastases | From treatment until end of study
  Data concerning the possible occurence of distant metastases will be collected from each patient from inclusion until end of study or date of death (an expected average time frame of 10 years).
Dyspnea | From inclusion until end of study
  From each included patient, dyspnea scores will be collected from start of treatment until end of study or date of death (an expected average time frame of 10 years).
Dysphagia | From treatment until end of study
  Dysphagia scores will be collected from each participating patient from treatment until end of study or date of death (an average time frame of 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Dekker, Dr, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands